CLINICAL TRIAL: NCT05531344
Title: Clinical Study of Composite Steep-pulse(High-frequency Irreversible Electroporation) Treatment Device Used in Patients With Benign Prostatic Hyperplasia
Brief Title: Composite Steep-pulseTreatment Device Used in Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: REMD Medical Technology (Industry)
Collaborators: RenJi Hospital (Other); Dongfang Hospital Affiliated to Tongji University (Other); Shanghai Pudong Hospital (Other); Qilu Hospital of Shandong University (Other); Ningbo No.2 Hospital (Other); Shangdong Yiyuan Hospital (Unknown); Tongji Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMD02
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: IRE; Composite Steep-pulse Treatment Device; Benign Prostatic Hyperplasia; randomized; medication-control; superiority; multi-center
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Composite Steep-pulse Treatment Device (Experimental): Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Device
  Interventions: Device: Composite Steep-pulse Treatment Device
- Tamsulosin (Active Comparator): Tamsulosin Hydrochloride Sustained Release Capsules, 0.2mg, once a day,3 months
  Interventions: Drug: Tamsulosin Hydrochloride Capsules

INTERVENTIONS:
Device: Composite Steep-pulse Treatment Device — Applying the Composite Steep-pulse Treatment Device to treat the patients with Benign Prostatic Hyperplasia
  Arms: Composite Steep-pulse Treatment Device
Drug: Tamsulosin Hydrochloride Capsules — Applying Tamsulosin Hydrochloride Capsules to treat the patients with Benign Prostatic Hyperplasia
  Arms: Tamsulosin

SUMMARY:
This is a prospective, randomized, open-label, parallel-group, medication-control, superiority, multicenter clinical study trial.

This study is studying the effects and safety in treating patients from nine different centers with Benign prostatic hyperplasia, employing Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Apparatus. This device could cause cell irreversible electroporation, which leading necrosis of hyperplasia tissue cells. It also has the ability to prevent nerve,vessel, urethral and capsule unnecessary injury beside the ablation area. Composite Steep-pulse Treatment Apparatus will be used in patients who pass inclusion/exclusion criteria. Safety, quality of life, and urodynamic data analysis of each patient will be evaluated in each study patients.

DETAILED DESCRIPTION:
Background:

Benign prostatic hyperplasia (BPH) is a frequently-occurring disease in elderly males. The incidence of BPH is as high as 50% in males over 50 years old, while the incidence of BPH is as high as 80% in males over 80 years old.

Current treatments for benign prostatic hyperplasia include oral drug therapy and surgical treatment. Drug therapy mainly includes:1. 5-α reductase inhibitors, such as Finasteride, which can delay or reduce the prostate volume, but it is required for 3-6 months to take effect, and patients need prolonged maintenance therapy. And it is contraindicated in patients with abnormal liver function, because the drug needs to be metabolized by the liver; 2. α receptor blockers, such as Tamsulosin and Doxazosin, which are able to relax the bladder neck, prostate and urethral smooth muscle, thereby reducing prostatic urethral resistance. It cannot reduce the size of the prostate gland, so it cannot fundamentally prevent the development of benign prostatic hyperplasia, while the effect on large volume benign prostatic hyperplasia is not obvious, and it is contraindicated in patients with renal insufficiency; 3 Traditional medicines, which can only be used as a supplementary drug.

Surgery is the second-line treatment of BPH, and its standard procedure is transurethral resection of the prostate (TURP), which is considered to be the gold standard surgical procedure due to its exact efficacy and minimally invasive nature. However, large-scale retrospective studies have shown severe complications after TURP, especially TURP syndrome, postoperative urinary incontinence, urethral stricture, etc., hence there are still many concerns about the application of this procedure. Although plasma transurethral resection of the prostate and various laser prostate surgeries have sprung up in recent years, the basic surgical operation concept is not changed and the common problems existing in the procedure cannot be completely avoided. Luckily, with the development of technology, more and more new and effective treatments have emerged for BPH.

In 2004, a new method using steep pulses to treat tumor was appeared. It showed that steep pulses could bring about Irreversible Electroporation (IRE) of cell, leading to necrosis of tumor or diseased cells. And it seemed to do no harms to the nerve and Vascular epithelial cell. The device of steep pulse had already been approved by FDA in 2011.However, this device of steep pulse has disadvantages like: (1)sever muscle contraction;(2)Urethral injury; (3)Capsule injury;(4)Nerve degeneration. This new device which is called Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Device, may have the potential to conquer these disadvantages.

Purpose:

1. This study will assess the efficacy of Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Device in the treatment of BPH.
2. This study will assess the safety of Composite Steep-pulse(High-frequency irreversible electroporation) Treatment Device in the treatment of BPH.

Methods:

1. patients recruitment
2. Irreversible Electroporation of malignant diseased Cell under Composite Steep-pulse Treatment for the patients with Benign Prostatic Hyperplasia;
3. Some factors such as prostate MRI, IPSS score, Qmax will be performed to evaluate the efficacy of the treatment.
4. Other factors such as the routine blood test, the routine urine test, the blood biochemistry test, ect. will be performed to evaluate the safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males between 50 to 80 years old;
2. Patients who Fully understand the treatment plan for irreversible electroporation, and accept the trial treatment and signed informed consent form;
3. International Prostate Symptom Score (IPSS)≥12;
4. Patients who have no willing to perform enucleation or transurethral resection of prostate;
5. Maximum urinary flow rate (Qmax) >5ml/min and ≤15ml/min, voided volume ≥150ml;
6. The volume of prostate was ≥30cm3 measured by MRI;
7. Patients who Could perform follow-up evaluation in accordance with the trial protocol.

Exclusion Criteria:

1. Patients with a history of prostate cancer, or who confirmed diagnosis of prostate cancer (needle biopsy of the prostate is required for patients indicated for needle aspiration, and if the needle result suggests benign prostatic hyperplasia, enrollment is allowed);
2. Patients with second-degree or higher atrioventricular block and other cardiac diseases with clear contraindications to anesthesia;
3. Patients with cardiac pacemakers and metallic replacement of pelvis or hip joints;
4. Patients who underwent previous prostate surgery for benign prostatic hyperplasia;
5. patients who have history of soft or rigid cystoscopy or other transurethral device use within 7 days prior to Informed Consent Form signed;
6. Any condition other than BPH that could lead to urinary symptoms or altered urinary flow rate (such as neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, acute or chronic urinary tract infection) as judged by the investigator;
7. Patients with a previous history of epilepsy;
8. Patients who have participated in other clinical trials within 3 months.
9. Patients with ASA (American Society of Anesthesiology) score 4 or above, such as malignant hypertension, recent myocardial infarction, active cerebrovascular accident, severe anemia and other contraindications to general anesthesia;
10. Patients who are considered to be inappropriate for participation in the trial by the investigator.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Difference value in urinary Qmax between 3 months after treatment with baseline. | 0,3 months
  The Qmax was measured before treatment, 1 month and 3 months after treatment,and baseline difference values (posttreatment-Pretreatment) were calculated. The difference value of Qmax at 3 months after treatment with baseline was used as the primary outcome.

SECONDARY OUTCOMES:
Difference value of size of prostate between different visits | 0,3 months
  Before and 3 months after treatment, prostate size was measured by prostate magnetic resonance scanning, and the rate of change was calculated.
Difference value of Qmax between different visits | 0,1,3 months
  Qmax was measured before treatment, 1 month and 3 months after treatment.
Difference value of IPSS score between different visits | 0,1,3 months
  Before treatment, 1 month and 3 months after treatment, the prostate function of the subjects was calculated according to the International Prostate Symptom Score (I PSS), and the total score and improvement score were counted, respectively.
Operability of host system of device | The day of surgery
  Evaluate the operability of the host system of device after surgery: satisfied, commonly, dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Remd Medical Technology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roehrborn CG, Siami P, Barkin J, Damiao R, Major-Walker K, Morrill B, Montorsi F; CombAT Study Group. The effects of dutasteride, tamsulosin and combination therapy on lower urinary tract symptoms in men with benign prostatic hyperplasia and prostatic enlargement: 2-year results from the CombAT study. J Urol. 2008 Feb;179(2):616-21; discussion 621. doi: 10.1016/j.juro.2007.09.084. Epub 2007 Dec 21. PMID 18082216